CLINICAL TRIAL: NCT05664672
Title: A Randomized, Controlled, Open-label Short-term Study to Evaluate Changes in Exposure to Harmful and Potentially Harmful Constituents in Adult Smokers Who Completely Switch to on!® Nicotine Pouches in a Clinical Setting
Brief Title: Study to Evaluate Changes in Smokers Using on!® Nicotine Pouches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altria Client Services LLC (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ALCS-REG-20-15-OTDN
Record Dates: First submitted 2022-12-16; First posted 2022-12-27 (Actual); Results first posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-10

CONDITIONS: Tobacco Use
Keywords: Tobacco; Smoking
MeSH Terms: conditions — Tobacco Use; Smoking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Group 1 (CC) (No Intervention): Subjects will be asked to continue smoking their UBCs ad libitum for 7 days.
- Group 2 (NP2) (Experimental): Subjects will exclusively use 2 mg NP, using at least 3 pouches per day for 7 days.
  Interventions: Other: OTDN Product 1
- Group 3 (NP4) (Experimental): Subjects will exclusively use 4 mg NP, using at least 3 pouches per day for 7 days.
  Interventions: Other: OTDN Product 2
- Group 4 (NP8) (Experimental): Subjects will exclusively use 8 mg NP, using at least 3 pouches per day for 7 days.
  Interventions: Other: OTDN Product 3
- Group 5 (NT) (Experimental): Subjects will completely stop all tobacco product usage for 7 days.
  Interventions: Other: No Tobacco

INTERVENTIONS:
Other: OTDN Product 1 — Mint on!® 2 mg nicotine pouches
  Arms: Group 2 (NP2)
Other: OTDN Product 2 — Mint on!® 4 mg nicotine pouches
  Arms: Group 3 (NP4)
Other: OTDN Product 3 — Mint on!® 8 mg nicotine pouches
  Arms: Group 4 (NP8)
Other: No Tobacco — subjects completely stop all tobacco product usage for 7 days
  Arms: Group 5 (NT)

SUMMARY:
The purpose of this study is to generate evidence regarding the extent of reduction in exposure to selected HPHCs in adult smokers switching to on!® NPs. The study intends to determine changes in exposure to selected HPHCs by measuring biomarkers in adult smokers who completely switch from smoking to use of on!® NP compared to those who continue smoking cigarettes or stop using all tobacco products.

DETAILED DESCRIPTION:
This is an open-label, randomized, 5 parallel-group clinical study evaluating changes in exposure to selected harmful and potentially harmful constituents (HPHCs) and product use behavior in adult smokers who are randomly assigned to 1 of the 5 groups; continue smoking, partially or completely switch to oral tobacco-derived nicotine products, or stop using any tobacco products for 7 days.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary consent to participate in this study documented on the signed ICF
2. Smoking history (self-reported at screening) of an average of at least 10 but no more than 30 factory-manufactured combustible cigarettes (either menthol or non-menthol) daily for at least 12 months prior to screening. Brief periods (ie, up to 7 consecutive days) of non-smoking during the 3 months prior to screening (eg, due to illness or participation in a study where smoking was prohibited) will be permitted
3. Positive urine cotinine (≥ 500 ng/mL) at screening
4. Female subjects who are heterosexually active and of childbearing potential (eg, neither surgically sterile at least 6 months prior to check-in nor postmenopausal with amenorrhea for at least 12 months prior to check-in with follicle-stimulating hormone [FSH] levels consistent with postmenopausal status) must have been using one of the following forms of contraception for the time period indicated and agree to continue using it through completion of the study:

   * Hormonal (eg, oral, vaginal ring, transdermal patch, implant, injection) consistently for at least 3 months prior to check-in, double barrier (ie, condom with spermicide or diaphragm with spermicide) consistently for at least 4 weeks prior to check-in, an intrauterine device for at least 4 months prior to check-in
   * Exclusive partner who has been vasectomized for at least 6 months (inclusive) prior to check-in

   Female subjects of childbearing potential who are not currently engaging in heterosexual intercourse must agree to use one of the above methods of birth control through completion of study, in the event that they have heterosexual intercourse during the course of the study.
5. Female subjects who are of nonchildbearing potential must have undergone one of the following sterilization procedures at least 6 months prior to check-in:

   Hysteroscopic sterilization (including Essure® or similar nonsurgical sterilization procedures); bilateral tubal ligation or bilateral salpingectomy; hysterectomy; bilateral oophorectomy

   Or be postmenopausal with amenorrhea for at least 12 months prior to check-in and have FSH levels consistent with postmenopausal status
6. Willing to comply with the requirements of the study
7. Willing to use all 3 on!® NP after the Product Trial at check-in
8. Willing and able to abstain from cigarettes from Day 1 through the end of the study (EOS)
9. Healthy adult males and females, 21 to 65 years of age, inclusive at screening, with subjects aged 46 to 65 years being fully vaccinated for COVID-19 (SARS-CoV-2) at least 14 days before the screening visit.

Exclusion Criteria:

1. Use of any type of tobacco- or nicotine-containing products other than manufactured cigarettes (eg, e-vapor products, roll-your-own cigarettes, bidis, snuff, nicotine inhaler, pipe, cigar, chewing tobacco, nicotine patch, nicotine spray, nicotine lozenge, or nicotine gum) in the 7 days prior to check-in
2. Self-reported puffers (ie, adult smokers who draw smoke from the cigarette into the mouth and throat but do not inhale)
3. Planning to quit smoking in the next 30 days (from screening visit)
4. History or presence of clinically significant gastrointestinal, renal, hepatic, neurologic, hematologic, endocrine, oncologic, urologic, existing respiratory diseases, immunologic, psychiatric, lymphatic, or cardiovascular disease, or any other condition that, in the opinion of the investigator, would jeopardize the safety of the subject or impact the validity of the study results
5. Clinically significant abnormal findings on the vital signs, physical examination, medical history, electrocardiogram (ECG), or clinical laboratory results, in the opinion of the investigator
6. Positive test for human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C virus at screening
7. History or presence of any type of malignant tumors
8. Current evidence or any history of congestive heart failure
9. Diabetes mellitus (fasting glucose ≥126 mg/L [7 mmol/L]) that is not controlled by diet/exercise alone, in the opinion of the investigator
10. An acute illness (eg, upper respiratory infection, viral infection) requiring treatment with prescribed medicines within 2 weeks prior to check-in
11. Dentition that prevents subjects from using on!® NP products
12. Allergic to or cannot tolerate mint flavoring agents or phenylalanine
13. Any planned surgery from the time of screening through EOS
14. History of drug or alcohol abuse within 24 months prior to check-in
15. Fever (ie, body temperature >100.5°F) at screening or check-in. One recheck may be performed at the investigator's discretion
16. Body mass index greater than 40.0 kg/m2 or less than 18.0 kg/m2 at screening
17. Systolic blood pressure >150 mmHg and/or diastolic blood pressure > 90 mmHg at screening or check-in, measured after being seated for at least 5 minutes. One recheck may be performed at the investigator's discretion
18. Estimated creatinine clearance (by Cockcroft-Gault equation) < 80 mL/minute at screening
19. Serum alanine aminotransferase ≥1.5 times the upper limit of normal and/or aspartate aminotransferase ≥1.5 times the upper limit of normal at screening
20. Positive screen for alcohol (breath) or any of the following drugs of abuse (urine), regardless of the reason of use: amphetamines, methamphetamines, opiates, cannabinoids, or cocaine at screening or check-in
21. Female subjects who are pregnant (positive serum pregnancy test at screening or urine pregnancy test at check-in), lactating, or intend to become pregnant from screening through EOS
22. Use of prescription or over-the-counter bronchodilator medication (eg, inhaled or oral ß-agonists) within 12 months prior to check-in
23. Use of medications or foods known or are suspected to interact with cytochrome P450 2A6 (including, but not limited to, amiodarone, amlodipine, amobarbital, buprenorphine, clofibrate, clotrimazole, desipramine, disulfiram, entacapone, fenofibrate, isoniazid, grapefruit, ketoconazole, letrozole, methimazole, methoxsalen, metyrapone, miconazole, modafinil, orphenadrine, pentobarbital, phenobarbital, pilocarpine, primidone, propoxyphene, quinidine, rifampicin, rifampin, secobarbital, selegiline, sulconazole, tioconazole, tranylcypromine) within 14 days or 5 half-lives of the drug, whichever is longer, prior to check-in or during the study
24. Use of antibiotic treatment within 2 weeks prior to check-in
25. Plasma donation within 7 days prior to check-in
26. Donation of blood or blood products (with the exception of plasma as noted above), had significant blood loss, or received whole blood or a blood product transfusion within 56 days prior to check-in
27. Participation in a previous clinical study for an investigational drug, device, biologic, or a tobacco product within 30 days prior to check-in
28. Participation in 2 or more Altria Client Services (ALCS) studies within the past 12-month period prior to check-in
29. Subject or a first-degree relative (ie, parent, sibling, child, spouse/partner) is a current or former employee of the tobacco industry or a named party or class representative in litigation with any tobacco company
30. Subject or a first-degree relative (ie, parent, sibling, child, spouse/partner) is a current employee of the study site
31. Positive result for coronavirus disease (COVID)-19 (SARS-CoV-2) test at screening or check-in
32. One or more "yes" answers to any of the questions on the COVID-19 (SARS-CoV-2) screening questionnaire (provided by the study site) at screening or check-in.
33. Have been diagnosed with major depressive disorder or have a history of suicide attempt.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Not more than 60% of either gender
Enrollment: 149 (Actual)
Dates: Start 2021-05-11 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J Howitt, MD, Principal Investigator — QPS Holdings LLC; William Smith, MD, Principal Investigator — NOCCR; Mark Adams, MD, Principal Investigator — CKRA
Locations (3):
- United States (3):
  - CKRA, Lexington, Kentucky
  - QPS, Springfield, Missouri
  - NOCCR, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After screening, subjects who met eligibility criteria but were not needed once sample size objectives were met, were discontinued. The remaining subjects participated in a brief Product Use Trial to allow them to become accustomed to the products prior to randomization. Subjects who did not meet the randomization criteria after completing the Product Use Trial were discontinued; these subjects are included in the safety population but were not assigned to a study group.
Groups:
- Not Assigned: Only includes subjects that enrolled in the study but dropped prior to randomization. This group includes subjects who participated in the Product Trial Period but withdrew before randomization.
Period: Overall Study
Arm/Group | Not Assigned | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
Started | 3 | 29 | 28 | 30 | 30 | 29
Completed | 0 | 28 | 25 | 30 | 25 | 22
Not Completed | 3 | 1 | 3 | 0 | 5 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 3 | 0 | 5 | 6
Not completed — Failure to Meet Randomization Criteria | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Met Eligibility Criteria But Not Needed | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population includes all subjects randomized to a study group (Group 1, 2, 3, 4 or 5), and any subject who was enrolled in the study but failed to meet randomization criteria and was discontinued by the PI. Subjects who met eligibility requirements but were not needed for the study are not included in the Baseline Analysis Population.
Groups:
- Not Assigned: Only include subjects that enrolled in the study but dropped prior to randomization. This group includes subjects who participated in the Product Trial Period but withdrew before randomization.
- Total: Total of all reporting groups
Arm/Group | Not Assigned | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT) | Total
Number analyzed (Participants) | 2 | 29 | 28 | 30 | 30 | 29 | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.0 (12.73) | 34.2 (7.51) | 33.6 (6.73) | 35.9 (8.49) | 31.7 (6.53) | 35.5 (7.29) | 34.2 (7.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 13 | 12 | 13 | 13 | 12 | 64
  Male | 1 | 16 | 16 | 17 | 17 | 17 | 84
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 2 | 28 | 27 | 30 | 30 | 28 | 145
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 8 | 7 | 13 | 16 | 10 | 54
  White | 2 | 21 | 20 | 17 | 14 | 17 | 91
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Height (cm) [Mean (Standard Deviation); unit: cm] | 170.00 (11.314) | 171.41 (10.442) | 174.16 (9.357) | 173.42 (8.530) | 172.35 (10.216) | 172.32 (9.781) | 172.73 (9.600)
Body Weight (kg) [Mean (Standard Deviation); unit: kg] | 89.55 (14.213) | 88.67 (19.968) | 92.61 (21.949) | 91.28 (20.291) | 85.82 (19.027) | 88.74 (19.284) | 89.39 (19.971)
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 30.87 (0.813) | 30.05 (5.528) | 30.42 (6.242) | 30.35 (6.336) | 28.94 (6.077) | 29.80 (5.687) | 29.90 (5.925)
Cigarettes per Day [Mean (Standard Deviation); unit: Cigarettes per day] | 16.50 (4.950) | 16.03 (5.519) | 16.14 (5.848) | 16.23 (5.425) | 16.57 (6.372) | 16.69 (5.439) | 16.34 (5.660)
Years of Smoking [Mean (Standard Deviation); unit: years] | 10.00 (0) | 16.15 (9.228) | 15.98 (6.784) | 16.71 (10.495) | 14.27 (7.924) | 15.94 (8.304) | 15.80 (8.579)
Fagerström test - Total score [Mean (Standard Deviation); unit: points] — The Fagerström Test assesses an individual's dependence on nicotine. It consists of Yes/No and multiple choice questions where each response is assigned a value from 0 to 1 (for yes/no questions) or 0 to 3 (for multiple choice questions). Values are summed to yield a total score with a minimum score of 0 points and a maximum score of 10 points. The higher the total Fagerström score, the more intense is the subject's physical dependence on nicotine. Population: The Fagerström Test for Cigarette Dependence was completed on the morning of Day 1 before any study product use. Subjects in the 'Not Assigned' group were discontinued prior to administration of the Fagerström Test and, therefore, the 'Number Analyzed' for this group is '0'.
  points
    number analyzed (Participants) | 0 | 29 | 28 | 30 | 30 | 29 | 146
    (all) |  | 4.7 (1.37) | 4.5 (1.71) | 5.1 (2.12) | 4.4 (1.92) | 5.4 (1.84) | 4.8 (1.83)

OUTCOME MEASURES:

1. Primary Outcome: NNAL Exposure in Subjects Using Nicotine Pouches for 7 Days Versus Subjects Who Continue to Smoke Cigarettes for 7 Days
Description: Summary of 24-hour urinary creatinine-adjusted total 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL) in subjects using nicotine pouches (NP) for 7 days versus subjects who continue to smoke cigarettes for 7 days and subjects who stopped using any tobacco products for 7 days.
  Total urine weight (g) collected during 24 hours was converted to 24-hour urine volume using assumed density of 1 g = 1 mL
  Amount of biomarker was calculated as:
  Urine Biomarker (unit2/24 hours) = Urine biomarker concentration [unit1/mL] × 24h urine volume [mL] ÷ 1000, where: unit2 = ng if unit1 = pg; unit2 = μg if unit1 = ng
  Adjusted Urine biomarker (unit2/g creatinine) = Urine biomarker concentration (unit1/mL) × 100 / Creatinine concentration (mg/dL), where unit2 = ng if unit1 = pg, and unit2 = μg if unit 1 = ng
  The absolute change from baseline of urine biomarker amount excreted in 24 hours was calculated as follows:
  Absolute change from baseline = Post Randomization Value - Baseline Value
Time Frame: Samples collected over 24 hours on Day -1 (baseline) and Day 7
Population: Biomarker of Exposure Population (BOE): All subjects from Groups 1, 2, 3, and 4 who used at least 1 of the assigned study products and all Group 5 subjects. To be included in the BOE population, subjects must have baseline (Day -1) and at least one post-baseline evaluable BOE data.
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
Number analyzed (Participants) | 28 | 22 | 30 | 25 | 21
ng/g
  Day -1 (Baseline) | 363 (239) | 274 (203) | 312 (201) | 293 (213) | 392 (308)
  Day 7 | 330 (224) | 67.8 (70.0) | 73.2 (42.7) | 64.7 (51.0) | 71.3 (62.2)
  Change from Baseline to Day 7 | -32.8 (67.6) | -206 (146) | -239 (172) | -228 (171) | -321 (290)
Statistical Analysis 1: Comparison: Group 1 (CC) vs Group 2 (NP2); Test type: Superiority; p < .0001, ANCOVA; Least square means (LSM) calculated from mixed model to control for variables were used for analysis instead of the observed means reported on table; Ratio of geometric LS means (Test/Ref) = 24.2, 95% CI 2-sided [15.9 to 37.0] — Geometric LSM calculated by transforming the natural-log LS means back to the linear scale. Ratio of geometric LSM expressed as percentage. In statistical model, group & gender included as fixed effects; baseline value included as covariate
Statistical Analysis 2: Comparison: Group 1 (CC) vs Group 3 (NP4); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 25.3, 95% CI 2-sided [17.1 to 37.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 1 (CC) vs Group 4 (NP8); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 22.4, 95% CI 2-sided [14.9 to 33.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1 (CC) vs Group 5 (NT); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 16.5, 95% CI 2-sided [10.8 to 25.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2 (NP2) vs Group 5 (NT); Test type: Superiority; p = 0.1148, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 147, 95% CI 2-sided [93.7 to 230] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3 (NP4) vs Group 5 (NT); Test type: Superiority; p = 0.0440, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 153, 95% CI 2-sided [101 to 233] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 4 (NP8) vs Group 5 (NT); Test type: Superiority; p = 0.2422, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 136, 95% CI 2-sided [87.8 to 210] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: NE Exposure in Subjects Using Nicotine Pouches for 7 Days Versus Subjects Who Continue to Smoke Cigarettes for 7 Days
Description: Summary of 24-hour urinary creatinine-adjusted Nicotine Equivalents (NE) in subjects using nicotine pouches (NP) for 7 days versus subjects who continue to smoke cigarettes for 7 days and subjects who stopped using any tobacco products for 7 days.
  Total urine weight (g) collected during the 24 hours was converted to 24-hour urine volume using the assumed density of 1 gram (g) equals 1 milliliter (mL).
  The amount of biomarker was calculated as follows:
  NE concentration (μg/mL) = (nicotine [ng/mL]/162.23 [mg/mmol] + nicotine-gluc [ng/mL]/338.36 [mg/mmol] + cotinine [ng/mL]/176.22 [mg/mmol] + cotinine-gluc [ng/mL]/352.34 [mg/mmol] + trans-3'-hydroxycotinine [ng/mL]/192.22 [mg/mmol] + trans-3'-hydroxycotinine-gluc [ng/mL]/368.34 [mg/mmol]) × 162.23 (mg/mmol) × 1 μg/1000 ng
  Adjusted Nicotine equivalents (mg NE/g creatinine) = NE concentration (μg/mL) × 100 / Creatinine concentration (mg/dL)
  Absolute change from baseline = Post Randomization Value - Baseline Value
Time Frame: Samples collected over 24 hours on Day -1 (baseline) and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
Number analyzed (Participants) | 28 | 22 | 30 | 25 | 21
mg/g
  Day -1 (Baseline) | 11.6 (6.55) | 8.73 (4.42) | 10.3 (4.83) | 10.5 (5.99) | 12.2 (7.34)
  Day 7 | 10.4 (5.10) | 5.79 (5.01) | 8.80 (6.66) | 11.8 (8.45) | 0.978 (2.35)
  Change from Baseline to Day 7 | -1.20 (3.81) | -2.94 (3.80) | -1.50 (5.81) | 1.34 (6.77) | -11.2 (6.89)
Statistical Analysis 1: Comparison: Group 1 (CC) vs Group 2 (NP2); Test type: Superiority; p = 0.0994, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 49.9, 95% CI 2-sided [22.7 to 110] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 1 (CC) vs Group 3 (NP4); Test type: Superiority; p = 0.4162, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 65.8, 95% CI 2-sided [32.0 to 135] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 1 (CC) vs Group 4 (NP8); Test type: Superiority; p = 1.0000, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 101, 95% CI 2-sided [47.5 to 215] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1 (CC) vs Group 5 (NT); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 2.23, 95% CI 2-sided [1.01 to 4.94] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2 (NP2) vs Group 5 (NT); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 2230, 95% CI 2-sided [965 to 5160] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3 (NP4) vs Group 5 (NT); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 2940, 95% CI 2-sided [1350 to 6400] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 4 (NP8) vs Group 5 (NT); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 4530, 95% CI 2-sided [2020 to 10200] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: 2-AN Exposure in Subjects Using Nicotine Pouches for 7 Days Versus Subjects Who Continue to Smoke Cigarettes for 7 Days
Description: Summary of 24-hour urinary creatinine-adjusted 2-aminonaphthalene (2-AN) in subjects using nicotine pouches (NP) for 7 days versus subjects who continue to smoke cigarettes for 7 days and subjects who stopped using any tobacco products for 7 days.
  Total urine weight (g) collected during 24 hours was converted to 24-hour urine volume using assumed density of 1 g = 1 mL
  Amount of biomarker was calculated as:
  Urine Biomarker (unit2/24 hours) = Urine biomarker concentration [unit1/mL] × 24h urine volume [mL] ÷ 1000, where: unit2 = ng if unit1 = pg; unit2 = μg if unit1 = ng
  Adjusted Urine biomarker (unit2/g creatinine) = Urine biomarker concentration (unit1/mL) × 100 / Creatinine concentration (mg/dL), where unit2 = ng if unit1 = pg, and unit2 = μg if unit 1 = ng
  The absolute change from baseline of urine biomarker amount excreted in 24 hours was calculated as follows:
  Absolute change from baseline = Post Randomization Value - Baseline Value
Time Frame: Samples collected over 24 hours on Day -1 (baseline) and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
Number analyzed (Participants) | 28 | 22 | 30 | 25 | 21
ng/g
  Day -1 (Baseline) | 21.7 (11.5) | 17.0 (9.93) | 21.6 (12.0) | 19.8 (11.2) | 20.6 (11.7)
  Day 7 | 20.2 (11.3) | 1.07 (0.728) | 1.82 (1.36) | 1.45 (1.35) | 1.29 (1.01)
  Change from Baseline to Day 7 | -1.58 (5.10) | -16.0 (9.77) | -19.8 (11.8) | -18.3 (10.9) | -19.3 (11.7)
Statistical Analysis 1: Comparison: Group 1 (CC) vs Group 2 (NP2); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 5.69, 95% CI 2-sided [3.29 to 9.87] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 1 (CC) vs Group 3 (NP4); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 8.08, 95% CI 2-sided [4.88 to 13.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 1 (CC) vs Group 4 (NP8); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 6.58, 95% CI 2-sided [3.88 to 11.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1 (CC) vs Group 5 (NT); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 6.03, 95% CI 2-sided [3.46 to 10.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2 (NP2) vs Group 5 (NT); Test type: Superiority; p = 0.9972, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 94.4, 95% CI 2-sided [52.7 to 169] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3 (NP4) vs Group 5 (NT); Test type: Superiority; p = 0.4655, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 134, 95% CI 2-sided [77.9 to 230] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 4 (NP8) vs Group 5 (NT); Test type: Superiority; p = 0.9851, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 109, 95% CI 2-sided [62.1 to 192] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: 4-ABP Exposure in Subjects Using Nicotine Pouches for 7 Days Versus Subjects Who Continue to Smoke Cigarettes for 7 Days
Description: Summary of 24-hour urinary creatinine-adjusted 4-aminobiphenyl (4-ABP) in subjects using nicotine pouches (NP) for 7 days versus subjects who continue to smoke cigarettes for 7 days and subjects who stopped using any tobacco products for 7 days.
  Total urine weight (g) collected during 24 hours was converted to 24-hour urine volume using assumed density of 1 g = 1 mL
  Amount of biomarker was calculated as:
  Urine Biomarker (unit2/24 hours) = Urine biomarker concentration [unit1/mL] × 24h urine volume [mL] ÷ 1000, where: unit2 = ng if unit1 = pg; unit2 = μg if unit1 = ng
  Adjusted Urine biomarker (unit2/g creatinine) = Urine biomarker concentration (unit1/mL) × 100 / Creatinine concentration (mg/dL), where unit2 = ng if unit1 = pg, and unit2 = μg if unit 1 = ng
  The absolute change from baseline of urine biomarker amount excreted in 24 hours was calculated as follows:
  Absolute change from baseline = Post Randomization Value - Baseline Value
Time Frame: Samples collected over 24 hours on Day -1 (baseline) and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
Number analyzed (Participants) | 28 | 22 | 30 | 25 | 21
ng/g
  Day -1 (Baseline) | 13.8 (6.74) | 10.2 (5.04) | 13.3 (6.29) | 12.8 (6.22) | 12.8 (6.81)
  Day 7 | 13.2 (7.44) | 1.42 (0.450) | 1.97 (0.749) | 1.72 (0.985) | 1.92 (1.04)
  Change from Baseline to Day 7 | -0.589 (4.53) | -8.75 (4.94) | -11.3 (6.04) | -11.1 (5.81) | -10.9 (6.58)
Statistical Analysis 1: Comparison: Group 1 (CC) vs Group 2 (NP2); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 13.7, 95% CI 2-sided [9.72 to 19.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 1 (CC) vs Group 3 (NP4); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 16.6, 95% CI 2-sided [12.1 to 22.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 1 (CC) vs Group 4 (NP8); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 13.4, 95% CI 2-sided [9.68 to 18.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1 (CC) vs Group 5 (NT); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 15.7, 95% CI 2-sided [11.2 to 22.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2 (NP2) vs Group 5 (NT); Test type: Superiority; p = 0.7167, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 86.8, 95% CI 2-sided [60.6 to 124] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3 (NP4) vs Group 5 (NT); Test type: Superiority; p = 0.9864, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 105, 95% CI 2-sided [75.3 to 147] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 4 (NP8) vs Group 5 (NT); Test type: Superiority; p = 0.5911, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 85.1, 95% CI 2-sided [60.1 to 120] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: HEMA Exposure in Subjects Using Nicotine Pouches for 7 Days Versus Subjects Who Continue to Smoke Cigarettes for 7 Days
Description: Summary of 24-hour urinary creatinine-adjusted 2-hydroxyethylmercapturic acid (HEMA) in subjects using nicotine pouches (NP) for 7 days versus subjects who continue to smoke cigarettes for 7 days and subjects who stopped using any tobacco products for 7 days.
  Total urine weight (g) collected during 24 hours was converted to 24-hour urine volume using assumed density of 1 g = 1 mL
  Amount of biomarker was calculated as:
  Urine Biomarker (unit2/24 hours) = Urine biomarker concentration [unit1/mL] × 24h urine volume [mL] ÷ 1000, where: unit2 = ng if unit1 = pg; unit2 = μg if unit1 = ng
  Adjusted Urine biomarker (unit2/g creatinine) = Urine biomarker concentration (unit1/mL) × 100 / Creatinine concentration (mg/dL), where unit2 = ng if unit1 = pg, and unit2 = μg if unit 1 = ng
  The absolute change from baseline of urine biomarker amount excreted in 24 hours was calculated as follows:
  Absolute change from baseline = Post Randomization Value - Baseline Value
Time Frame: Samples collected over 24 hours on Day -1 (baseline) and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
Number analyzed (Participants) | 28 | 22 | 30 | 25 | 21
μg/g
  Day -1 (Baseline) | 5.19 (5.34) | 2.98 (1.69) | 5.64 (5.29) | 5.65 (6.11) | 3.90 (3.42)
  Day 7 | 4.63 (4.47) | 0.959 (0.660) | 1.18 (0.758) | 1.55 (1.11) | 1.30 (0.762)
  Change from Baseline to Day 7 | -0.559 (1.80) | -2.03 (1.40) | -4.46 (4.63) | -4.09 (5.50) | -2.60 (3.22)
Statistical Analysis 1: Comparison: Group 1 (CC) vs Group 2 (NP2); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 29.6, 95% CI 2-sided [21.8 to 40.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 1 (CC) vs Group 3 (NP4); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 28.3, 95% CI 2-sided [21.5 to 37.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 1 (CC) vs Group 4 (NP8); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 33.1, 95% CI 2-sided [24.8 to 44.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1 (CC) vs Group 5 (NT); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 37.5, 95% CI 2-sided [27.7 to 50.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2 (NP2) vs Group 5 (NT); Test type: Superiority; p = 0.1950, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 78.8, 95% CI 2-sided [57.3 to 108] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3 (NP4) vs Group 5 (NT); Test type: Superiority; p = 0.0699, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 75.5, 95% CI 2-sided [56.1 to 102] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 4 (NP8) vs Group 5 (NT); Test type: Superiority; p = 0.7041, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 88.3, 95% CI 2-sided [64.7 to 120] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: CEMA Exposure in Subjects Using Nicotine Pouches for 7 Days Versus Subjects Who Continue to Smoke Cigarettes for 7 Days
Description: Summary of 24-hour urinary creatinine-adjusted cyanoethylmercapturic acid (CEMA) in subjects using nicotine pouches (NP) for 7 days versus subjects who continue to smoke cigarettes for 7 days and subjects who stopped using any tobacco products for 7 days.
  Total urine weight (g) collected during 24 hours was converted to 24-hour urine volume using assumed density of 1 g = 1 mL
  Amount of biomarker was calculated as:
  Urine Biomarker (unit2/24 hours) = Urine biomarker concentration [unit1/mL] × 24h urine volume [mL] ÷ 1000, where: unit2 = ng if unit1 = pg; unit2 = μg if unit1 = ng
  Adjusted Urine biomarker (unit2/g creatinine) = Urine biomarker concentration (unit1/mL) × 100 / Creatinine concentration (mg/dL), where unit2 = ng if unit1 = pg, and unit2 = μg if unit 1 = ng
  The absolute change from baseline of urine biomarker amount excreted in 24 hours was calculated as follows:
  Absolute change from baseline = Post Randomization Value - Baseline Value
Time Frame: Samples collected over 24 hours on Day -1 (baseline) and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
Number analyzed (Participants) | 28 | 22 | 30 | 25 | 21
μg/g
  Day -1 (Baseline) | 163 (74.1) | 133 (65.0) | 154 (83.4) | 170 (72.9) | 160 (94.8)
  Day 7 | 150 (72.1) | 17.4 (10.3) | 18.9 (10.7) | 23.0 (13.1) | 16.0 (11.6)
  Change from Baseline to Day 7 | -12.4 (28.9) | -116 (56.6) | -135 (75.8) | -147 (67.5) | -144 (85.4)
Statistical Analysis 1: Comparison: Group 1 (CC) vs Group 2 (NP2); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 13.3, 95% CI 2-sided [9.57 to 18.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 1 (CC) vs Group 3 (NP4); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 13.3, 95% CI 2-sided [9.84 to 17.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 1 (CC) vs Group 4 (NP8); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 13.6, 95% CI 2-sided [9.93 to 18.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1 (CC) vs Group 5 (NT); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 9.28, 95% CI 2-sided [6.67 to 12.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2 (NP2) vs Group 5 (NT); Test type: Superiority; p = 0.0404, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 143, 95% CI 2-sided [101 to 202] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3 (NP4) vs Group 5 (NT); Test type: Superiority; p = 0.0243, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 143, 95% CI 2-sided [104 to 198] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 4 (NP8) vs Group 5 (NT); Test type: Superiority; p = 0.0215, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 146, 95% CI 2-sided [105 to 205] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: SPMA Exposure in Subjects Using Nicotine Pouches for 7 Days Versus Subjects Who Continue to Smoke Cigarettes for 7 Days
Description: Summary of 24-hour urinary creatinine-adjusted S-phenylmercapturic acid (SPMA) in subjects using nicotine pouches (NP) for 7 days versus subjects who continue to smoke cigarettes for 7 days and subjects who stopped using any tobacco products for 7 days.
  Total urine weight (g) collected during 24 hours was converted to 24-hour urine volume using assumed density of 1 g = 1 mL
  Amount of biomarker was calculated as:
  Urine Biomarker (unit2/24 hours) = Urine biomarker concentration [unit1/mL] × 24h urine volume [mL] ÷ 1000, where: unit2 = ng if unit1 = pg; unit2 = μg if unit1 = ng
  Adjusted Urine biomarker (unit2/g creatinine) = Urine biomarker concentration (unit1/mL) × 100 / Creatinine concentration (mg/dL), where unit2 = ng if unit1 = pg, and unit2 = μg if unit 1 = ng
  The absolute change from baseline of urine biomarker amount excreted in 24 hours was calculated as follows:
  Absolute change from baseline = Post Randomization Value - Baseline Value
Time Frame: Samples collected over 24 hours on Day -1 (baseline) and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
Number analyzed (Participants) | 28 | 22 | 30 | 25 | 21
μg/g
  Day -1 (Baseline) | 4.41 (3.29) | 3.03 (2.24) | 3.90 (2.41) | 3.79 (2.70) | 3.54 (3.18)
  Day 7 | 4.14 (3.24) | 0.149 (0.108) | 0.183 (0.106) | 0.186 (0.140) | 0.171 (0.107)
  Change from Baseline to Day 7 | -0.265 (0.810) | -2.88 (2.17) | -3.72 (2.38) | -3.61 (2.67) | -3.37 (3.09)
Statistical Analysis 1: Comparison: Group 1 (CC) vs Group 2 (NP2); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 5.37, 95% CI 2-sided [3.69 to 7.80] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 1 (CC) vs Group 3 (NP4); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 5.65, 95% CI 2-sided [4.01 to 7.96] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 1 (CC) vs Group 4 (NP8); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 5.61, 95% CI 2-sided [3.92 to 8.03] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1 (CC) vs Group 5 (NT); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 6.09, 95% CI 2-sided [4.17 to 8.89] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2 (NP2) vs Group 5 (NT); Test type: Superiority; p = 0.8335, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 88.1, 95% CI 2-sided [59.4 to 131] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3 (NP4) vs Group 5 (NT); Test type: Superiority; p = 0.9622, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 92.9, 95% CI 2-sided [64.2 to 134] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 4 (NP8) vs Group 5 (NT); Test type: Superiority; p = 0.9531, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 92.1, 95% CI 2-sided [62.8 to 135] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: HMPMA Exposure in Subjects Using Nicotine Pouches for 7 Days Versus Subjects Who Continue to Smoke Cigarettes for 7 Days
Description: Summary of 24-hour urinary creatinine-adjusted 3-hydroxy-1-methylpropylmercapturic acid (HMPMA) in subjects using nicotine pouches (NP) for 7 days versus subjects who continue to smoke cigarettes for 7 days and subjects who stopped using any tobacco products for 7 days.
  Total urine weight (g) collected during 24 hours was converted to 24-hour urine volume using assumed density of 1 g = 1 mL
  Amount of biomarker was calculated as:
  Urine Biomarker (unit2/24 hours) = Urine biomarker concentration [unit1/mL] × 24h urine volume [mL] ÷ 1000, where: unit2 = ng if unit1 = pg; unit2 = μg if unit1 = ng
  Adjusted Urine biomarker (unit2/g creatinine) = Urine biomarker concentration (unit1/mL) × 100 / Creatinine concentration (mg/dL), where unit2 = ng if unit1 = pg, and unit2 = μg if unit 1 = ng
  The absolute change from baseline of urine biomarker amount excreted in 24 hours was calculated as follows:
  Absolute change from baseline = Post Randomization Value - Baseline Value
Time Frame: Samples collected over 24 hours on Day -1 (baseline) and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
Number analyzed (Participants) | 28 | 22 | 30 | 25 | 21
μg/g
  Day -1 (Baseline) | 371 (161) | 303 (121) | 325 (167) | 338 (143) | 353 (198)
  Day 7 | 345 (159) | 53.4 (10.4) | 57.1 (25.0) | 48.6 (10.3) | 55.2 (12.4)
  Change from Baseline to Day 7 | -25.6 (75.6) | -250 (120) | -268 (163) | -290 (142) | -298 (197)
Statistical Analysis 1: Comparison: Group 1 (CC) vs Group 2 (NP2); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 18.0, 95% CI 2-sided [14.4 to 22.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 1 (CC) vs Group 3 (NP4); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 18.0, 95% CI 2-sided [14.8 to 22.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 1 (CC) vs Group 4 (NP8); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 15.8, 95% CI 2-sided [12.8 to 19.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1 (CC) vs Group 5 (NT); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 18.2, 95% CI 2-sided [14.6 to 22.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2 (NP2) vs Group 5 (NT); Test type: Superiority; p = 0.9993, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 98.4, 95% CI 2-sided [78.2 to 124] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3 (NP4) vs Group 5 (NT); Test type: Superiority; p = 0.9998, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 98.9, 95% CI 2-sided [79.7 to 123] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 4 (NP8) vs Group 5 (NT); Test type: Superiority; p = 0.3019, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 86.4, 95% CI 2-sided [69.1 to 108] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: 3-HPMA Exposure in Subjects Using Nicotine Pouches for 7 Days Versus Subjects Who Continue to Smoke Cigarettes for 7 Days
Description: Summary of 24-hour urinary creatinine-adjusted 3-hydroxypropylmercapturic acid (3-HPMA) in subjects using nicotine pouches (NP) for 7 days versus subjects who continue to smoke cigarettes for 7 days and subjects who stopped using any tobacco products for 7 days.
  Total urine weight (g) collected during 24 hours was converted to 24-hour urine volume using assumed density of 1 g = 1 mL
  Amount of biomarker was calculated as:
  Urine Biomarker (unit2/24 hours) = Urine biomarker concentration [unit1/mL] × 24h urine volume [mL] ÷ 1000, where: unit2 = ng if unit1 = pg; unit2 = μg if unit1 = ng
  Adjusted Urine biomarker (unit2/g creatinine) = Urine biomarker concentration (unit1/mL) × 100 / Creatinine concentration (mg/dL), where unit2 = ng if unit1 = pg, and unit2 = μg if unit 1 = ng
  The absolute change from baseline of urine biomarker amount excreted in 24 hours was calculated as follows:
  Absolute change from baseline = Post Randomization Value - Baseline Value
Time Frame: Samples collected over 24 hours on Day -1 (baseline) and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
Number analyzed (Participants) | 28 | 22 | 30 | 25 | 21
μg/g
  Day -1 (Baseline) | 1250 (605) | 969 (414) | 1160 (550) | 1170 (516) | 1200 (844)
  Day 7 | 1170 (614) | 195 (98.9) | 259 (118) | 215 (98.7) | 281 (205)
  Change from Baseline to Day 7 | -82.7 (299) | -774 (410) | -897 (557) | -957 (494) | -923 (836)
Statistical Analysis 1: Comparison: Group 1 (CC) vs Group 2 (NP2); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 18.3, 95% CI 2-sided [13.2 to 25.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 1 (CC) vs Group 3 (NP4); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 23.7, 95% CI 2-sided [17.6 to 31.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 1 (CC) vs Group 4 (NP8); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 19.3, 95% CI 2-sided [14.2 to 26.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1 (CC) vs Group 5 (NT); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 24.0, 95% CI 2-sided [17.3 to 33.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2 (NP2) vs Group 5 (NT); Test type: Superiority; p = 0.1530, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 76.1, 95% CI 2-sided [54.0 to 107] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3 (NP4) vs Group 5 (NT); Test type: Superiority; p = 0.9999, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 98.6, 95% CI 2-sided [71.7 to 136] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 4 (NP8) vs Group 5 (NT); Test type: Superiority; p = 0.3025, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 80.5, 95% CI 2-sided [57.8 to 112] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: 2-HPMA Exposure in Subjects Using Nicotine Pouches for 7 Days Versus Subjects Who Continue to Smoke Cigarettes for 7 Days
Description: Summary of 24-hour urinary creatinine-adjusted 2-hydroxypropylmercapturic acid (2-HPMA) in subjects using nicotine pouches (NP) for 7 days versus subjects who continue to smoke cigarettes for 7 days and subjects who stopped using any tobacco products for 7 days.
  Total urine weight (g) collected during 24 hours was converted to 24-hour urine volume using assumed density of 1 g = 1 mL
  Amount of biomarker was calculated as:
  Urine Biomarker (unit2/24 hours) = Urine biomarker concentration [unit1/mL] × 24h urine volume [mL] ÷ 1000, where: unit2 = ng if unit1 = pg; unit2 = μg if unit1 = ng
  Adjusted Urine biomarker (unit2/g creatinine) = Urine biomarker concentration (unit1/mL) × 100 / Creatinine concentration (mg/dL), where unit2 = ng if unit1 = pg, and unit2 = μg if unit 1 = ng
  The absolute change from baseline of urine biomarker amount excreted in 24 hours was calculated as follows:
  Absolute change from baseline = Post Randomization Value - Baseline Value
Time Frame: Samples collected over 24 hours on Day -1 (baseline) and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
Number analyzed (Participants) | 28 | 22 | 30 | 25 | 21
μg/g
  Day -1 (Baseline) | 52.7 (28.7) | 39.2 (19.4) | 47.3 (28.4) | 45.4 (23.8) | 41.4 (23.6)
  Day 7 | 50.9 (31.8) | 9.44 (3.87) | 11.9 (3.97) | 12.5 (7.43) | 11.9 (3.97)
  Change from Baseline to Day 7 | -1.81 (13.8) | -29.8 (20.4) | -35.4 (26.9) | -33.0 (26.0) | -29.6 (22.4)
Statistical Analysis 1: Comparison: Group 1 (CC) vs Group 2 (NP2); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 22.7, 95% CI 2-sided [17.0 to 30.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 1 (CC) vs Group 3 (NP4); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 28.1, 95% CI 2-sided [21.6 to 36.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 1 (CC) vs Group 4 (NP8); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 27.5, 95% CI 2-sided [20.8 to 36.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1 (CC) vs Group 5 (NT); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 28.7, 95% CI 2-sided [21.4 to 38.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2 (NP2) vs Group 5 (NT); Test type: Superiority; p = 0.1843, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 79.4, 95% CI 2-sided [58.6 to 108] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3 (NP4) vs Group 5 (NT); Test type: Superiority; p = 0.9994, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 98.1, 95% CI 2-sided [73.9 to 130] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 4 (NP8) vs Group 5 (NT); Test type: Superiority; p = 0.9891, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 95.9, 95% CI 2-sided [71.4 to 129] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: AAMA Exposure in Subjects Using Nicotine Pouches for 7 Days Versus Subjects Who Continue to Smoke Cigarettes for 7 Days
Description: Summary of 24-hour urinary creatinine-adjusted N-acetyl-S-(2-carbamoylethyl) cysteine (AAMA) in subjects using nicotine pouches (NP) for 7 days versus subjects who continue to smoke cigarettes for 7 days and subjects who stopped using any tobacco products for 7 days.
  Total urine weight (g) collected during 24 hours was converted to 24-hour urine volume using assumed density of 1 g = 1 mL
  Amount of biomarker was calculated as:
  Urine Biomarker (unit2/24 hours) = Urine biomarker concentration [unit1/mL] × 24h urine volume [mL] ÷ 1000, where: unit2 = ng if unit1 = pg; unit2 = μg if unit1 = ng
  Adjusted Urine biomarker (unit2/g creatinine) = Urine biomarker concentration (unit1/mL) × 100 / Creatinine concentration (mg/dL), where unit2 = ng if unit1 = pg, and unit2 = μg if unit 1 = ng
  The absolute change from baseline of urine biomarker amount excreted in 24 hours was calculated as follows:
  Absolute change from baseline = Post Randomization Value - Baseline Value
Time Frame: Samples collected over 24 hours on Day -1 (baseline) and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
Number analyzed (Participants) | 28 | 22 | 30 | 25 | 21
μg/g
  Day -1 (Baseline) | 92.6 (30.5) | 82.6 (36.1) | 95.6 (29.7) | 94.0 (36.4) | 94.3 (46.0)
  Day 7 | 87.7 (31.8) | 29.4 (6.96) | 39.1 (12.7) | 36.7 (13.4) | 35.9 (10.4)
  Change from Baseline to Day 7 | -4.90 (19.0) | -53.1 (33.0) | -56.5 (27.0) | -57.3 (32.1) | -58.3 (43.1)
Statistical Analysis 1: Comparison: Group 1 (CC) vs Group 2 (NP2); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 37.3, 95% CI 2-sided [30.4 to 45.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 1 (CC) vs Group 3 (NP4); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 44.0, 95% CI 2-sided [36.5 to 53.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 1 (CC) vs Group 4 (NP8); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 41.8, 95% CI 2-sided [34.4 to 50.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1 (CC) vs Group 5 (NT); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 42.9, 95% CI 2-sided [34.9 to 52.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2 (NP2) vs Group 5 (NT); Test type: Superiority; p = 0.3027, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 86.9, 95% CI 2-sided [70.0 to 108] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3 (NP4) vs Group 5 (NT); Test type: Superiority; p = 0.9926, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 103, 95% CI 2-sided [83.9 to 125] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 4 (NP8) vs Group 5 (NT); Test type: Superiority; p = 0.9938, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 97.5, 95% CI 2-sided [79.1 to 120] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: GAMA Exposure in Subjects Using Nicotine Pouches for 7 Days Versus Subjects Who Continue to Smoke Cigarettes for 7 Days
Description: Summary of 24-hour urinary creatinine-adjusted N-acetyl-S-(2-carbamoyl-2-hydroxyethyl)-1-cysteine (GAMA) in subjects using nicotine pouches (NP) for 7 days versus subjects who continue to smoke cigarettes for 7 days and subjects who stopped using any tobacco products for 7 days.
  Total urine weight (g) collected during 24 hours was converted to 24-hour urine volume using assumed density of 1 g = 1 mL
  Amount of biomarker was calculated as:
  Urine Biomarker (unit2/24 hours) = Urine biomarker concentration [unit1/mL] × 24h urine volume [mL] ÷ 1000, where: unit2 = ng if unit1 = pg; unit2 = μg if unit1 = ng
  Adjusted Urine biomarker (unit2/g creatinine) = Urine biomarker concentration (unit1/mL) × 100 / Creatinine concentration (mg/dL), where unit2 = ng if unit1 = pg, and unit2 = μg if unit 1 = ng
  The absolute change from baseline of urine biomarker amount excreted in 24 hours was calculated as follows:
  Absolute change from baseline = Post Randomization Value - Baseline Value
Time Frame: Samples collected over 24 hours on Day -1 (baseline) and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
Number analyzed (Participants) | 28 | 22 | 30 | 25 | 21
μg/g
  Day -1 (Baseline) | 14.4 (6.15) | 13.1 (5.27) | 14.3 (4.29) | 14.7 (5.23) | 14.1 (5.89)
  Day 7 | 14.1 (6.48) | 5.93 (1.94) | 7.58 (1.88) | 7.30 (2.24) | 7.26 (2.26)
  Change from Baseline to Day 7 | -0.256 (3.59) | -7.20 (3.99) | -6.77 (3.51) | -7.35 (4.11) | -6.79 (4.94)
Statistical Analysis 1: Comparison: Group 1 (CC) vs Group 2 (NP2); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 46.3, 95% CI 2-sided [39.5 to 54.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 1 (CC) vs Group 3 (NP4); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 55.6, 95% CI 2-sided [48.0 to 64.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 1 (CC) vs Group 4 (NP8); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 52.7, 95% CI 2-sided [45.2 to 61.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1 (CC) vs Group 5 (NT); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 54.9, 95% CI 2-sided [46.7 to 64.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2 (NP2) vs Group 5 (NT); Test type: Superiority; p = 0.0504, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 84.4, 95% CI 2-sided [71.2 to 100] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3 (NP4) vs Group 5 (NT); Test type: Superiority; p = 0.9988, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 101, 95% CI 2-sided [86.4 to 119] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 4 (NP8) vs Group 5 (NT); Test type: Superiority; p = 0.9238, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 96.0, 95% CI 2-sided [81.4 to 113] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: 2-MHBMA Exposure in Subjects Using Nicotine Pouches for 7 Days Versus Subjects Who Continue to Smoke Cigarettes for 7 Days
Description: Summary of 24-hour urinary creatinine-adjusted 2-hydroxybutenylmercapturic acid (2-MHBMA) in subjects using nicotine pouches (NP) for 7 days versus subjects who continue to smoke cigarettes for 7 days and subjects who stopped using any tobacco products for 7 days.
  Total urine weight (g) collected during 24 hours was converted to 24-hour urine volume using assumed density of 1 g = 1 mL
  Amount of biomarker was calculated as:
  Urine Biomarker (unit2/24 hours) = Urine biomarker concentration [unit1/mL] × 24h urine volume [mL] ÷ 1000, where: unit2 = ng if unit1 = pg; unit2 = μg if unit1 = ng
  Adjusted Urine biomarker (unit2/g creatinine) = Urine biomarker concentration (unit1/mL) × 100 / Creatinine concentration (mg/dL), where unit2 = ng if unit1 = pg, and unit2 = μg if unit 1 = ng
  The absolute change from baseline of urine biomarker amount excreted in 24 hours was calculated as follows:
  Absolute change from baseline = Post Randomization Value - Baseline Value
Time Frame: Samples collected over 24 hours on Day -1 (baseline) and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
Number analyzed (Participants) | 28 | 22 | 30 | 25 | 21
μg/g
  Day -1 (Baseline) | 1.93 (1.53) | 1.24 (1.12) | 1.60 (1.66) | 1.47 (1.37) | 1.26 (1.15)
  Day 7 | 1.74 (1.33) | 0.0359 (0.0338) | 0.0487 (0.0466) | 0.0460 (0.0413) | 0.0729 (0.0800)
  Change from Baseline to Day 7 | -0.194 (0.517) | -1.20 (1.11) | -1.56 (1.63) | -1.43 (1.36) | -1.19 (1.11)
Statistical Analysis 1: Comparison: Group 1 (CC) vs Group 2 (NP2); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 3.71, 95% CI 2-sided [1.88 to 7.31] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 1 (CC) vs Group 3 (NP4); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 4.25, 95% CI 2-sided [2.28 to 7.93] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 1 (CC) vs Group 4 (NP8); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 4.24, 95% CI 2-sided [2.20 to 8.14] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1 (CC) vs Group 5 (NT); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 6.40, 95% CI 2-sided [3.22 to 12.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2 (NP2) vs Group 5 (NT); Test type: Superiority; p = 0.1840, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 57.9, 95% CI 2-sided [28.3 to 119] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3 (NP4) vs Group 5 (NT); Test type: Superiority; p = 0.3552, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 66.4, 95% CI 2-sided [34.0 to 130] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 4 (NP8) vs Group 5 (NT); Test type: Superiority; p = 0.3810, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 66.2, 95% CI 2-sided [33.0 to 133] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: 2-OH-Flu Exposure in Subjects Using Nicotine Pouches for 7 Days Versus Subjects Who Continue to Smoke Cigarettes for 7 Days
Description: Summary of 24-hour urinary creatinine-adjusted 2-OH-Fluorene (2-OH-Flu) in subjects using nicotine pouches (NP) for 7 days versus subjects who continue to smoke cigarettes for 7 days and subjects who stopped using any tobacco products for 7 days.
  Total urine weight (g) collected during 24 hours was converted to 24-hour urine volume using assumed density of 1 g = 1 mL
  Amount of biomarker was calculated as:
  Urine Biomarker (unit2/24 hours) = Urine biomarker concentration [unit1/mL] × 24h urine volume [mL] ÷ 1000, where: unit2 = ng if unit1 = pg; unit2 = μg if unit1 = ng
  Adjusted Urine biomarker (unit2/g creatinine) = Urine biomarker concentration (unit1/mL) × 100 / Creatinine concentration (mg/dL), where unit2 = ng if unit1 = pg, and unit2 = μg if unit 1 = ng
  The absolute change from baseline of urine biomarker amount excreted in 24 hours was calculated as follows:
  Absolute change from baseline = Post Randomization Value - Baseline Value
Time Frame: Samples collected over 24 hours on Day -1 (baseline) and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
Number analyzed (Participants) | 28 | 22 | 30 | 25 | 21
μg/g
  Day -1 (Baseline) | 2.24 (1.11) | 1.71 (0.890) | 2.01 (1.08) | 2.14 (1.09) | 2.08 (1.11)
  Day 7 | 2.08 (1.17) | 0.280 (0.144) | 0.356 (0.141) | 0.361 (0.225) | 0.345 (0.203)
  Change from Baseline to Day 7 | -0.159 (0.401) | -1.43 (0.777) | -1.65 (0.995) | -1.78 (0.916) | -1.73 (0.931)
Statistical Analysis 1: Comparison: Group 1 (CC) vs Group 2 (NP2); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 16.8, 95% CI 2-sided [13.0 to 21.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 1 (CC) vs Group 3 (NP4); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 20.5, 95% CI 2-sided [16.2 to 25.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 1 (CC) vs Group 4 (NP8); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 18.2, 95% CI 2-sided [14.3 to 23.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1 (CC) vs Group 5 (NT); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 17.8, 95% CI 2-sided [13.7 to 23.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2 (NP2) vs Group 5 (NT); Test type: Superiority; p = 0.9589, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 94.5, 95% CI 2-sided [72.0 to 124] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3 (NP4) vs Group 5 (NT); Test type: Superiority; p = 0.4442, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 115, 95% CI 2-sided [89.3 to 148] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 4 (NP8) vs Group 5 (NT); Test type: Superiority; p = 0.9975, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 103, 95% CI 2-sided [78.8 to 133] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: 2-OH-Nap Exposure in Subjects Using Nicotine Pouches for 7 Days Versus Subjects Who Continue to Smoke Cigarettes for 7 Days
Description: Summary of 24-hour urinary creatinine-adjusted 2-Naphthol (2-OH-Nap) in subjects using nicotine pouches (NP) for 7 days versus subjects who continue to smoke cigarettes for 7 days and subjects who stopped using any tobacco products for 7 days.
  Total urine weight (g) collected during 24 hours was converted to 24-hour urine volume using assumed density of 1 g = 1 mL
  Amount of biomarker was calculated as:
  Urine Biomarker (unit2/24 hours) = Urine biomarker concentration [unit1/mL] × 24h urine volume [mL] ÷ 1000, where: unit2 = ng if unit1 = pg; unit2 = μg if unit1 = ng
  Adjusted Urine biomarker (unit2/g creatinine) = Urine biomarker concentration (unit1/mL) × 100 / Creatinine concentration (mg/dL), where unit2 = ng if unit1 = pg, and unit2 = μg if unit 1 = ng
  The absolute change from baseline of urine biomarker amount excreted in 24 hours was calculated as follows:
  Absolute change from baseline = Post Randomization Value - Baseline Value
Time Frame: Samples collected over 24 hours on Day -1 (baseline) and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
Number analyzed (Participants) | 28 | 22 | 30 | 25 | 21
μg/g
  Day -1 (Baseline) | 11.1 (5.08) | 11.5 (8.46) | 12.6 (5.56) | 13.8 (7.01) | 11.8 (7.60)
  Day 7 | 10.6 (5.06) | 5.16 (6.38) | 5.26 (3.89) | 4.80 (4.38) | 6.00 (5.56)
  Change from Baseline to Day 7 | -0.550 (2.55) | -6.38 (3.86) | -7.31 (5.20) | -9.00 (5.09) | -5.81 (5.91)
Statistical Analysis 1: Comparison: Group 1 (CC) vs Group 2 (NP2); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 36.5, 95% CI 2-sided [23.9 to 55.6] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 1 (CC) vs Group 3 (NP4); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 39.9, 95% CI 2-sided [27.1 to 59.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 1 (CC) vs Group 4 (NP8); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 30.2, 95% CI 2-sided [20.1 to 45.5] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1 (CC) vs Group 5 (NT); Test type: Superiority; p = 0.0002, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 48.9, 95% CI 2-sided [31.9 to 75.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2 (NP2) vs Group 5 (NT); Test type: Superiority; p = 0.2938, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 74.5, 95% CI 2-sided [47.6 to 117] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3 (NP4) vs Group 5 (NT); Test type: Superiority; p = 0.5552, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 81.6, 95% CI 2-sided [53.7 to 124] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 4 (NP8) vs Group 5 (NT); Test type: Superiority; p = 0.0254, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 61.7, 95% CI 2-sided [39.9 to 95.5] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: 1-OH-Phe Exposure in Subjects Using Nicotine Pouches for 7 Days Versus Subjects Who Continue to Smoke Cigarettes for 7 Days
Description: Summary of 24-hour urinary creatinine-adjusted 1-OH-Phenanthrene (1-OH-Phe) in subjects using nicotine pouches (NP) for 7 days versus subjects who continue to smoke cigarettes for 7 days and subjects who stopped using any tobacco products for 7 days.
  Total urine weight (g) collected during 24 hours was converted to 24-hour urine volume using assumed density of 1 g = 1 mL
  Amount of biomarker was calculated as:
  Urine Biomarker (unit2/24 hours) = Urine biomarker concentration [unit1/mL] × 24h urine volume [mL] ÷ 1000, where: unit2 = ng if unit1 = pg; unit2 = μg if unit1 = ng
  Adjusted Urine biomarker (unit2/g creatinine) = Urine biomarker concentration (unit1/mL) × 100 / Creatinine concentration (mg/dL), where unit2 = ng if unit1 = pg, and unit2 = μg if unit 1 = ng
  The absolute change from baseline of urine biomarker amount excreted in 24 hours was calculated as follows:
  Absolute change from baseline = Post Randomization Value - Baseline Value
Time Frame: Samples collected over 24 hours on Day -1 (baseline) and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
Number analyzed (Participants) | 28 | 22 | 30 | 25 | 21
μg/g
  Day -1 (Baseline) | 0.218 (0.107) | 0.162 (0.0816) | 0.172 (0.0938) | 0.171 (0.0902) | 0.191 (0.0895)
  Day 7 | 0.203 (0.108) | 0.0804 (0.0397) | 0.0804 (0.0397) | 0.0674 (0.0380) | 0.0833 (0.0431)
  Change from Baseline to Day 7 | -0.0142 (0.0517) | -0.0818 (0.0592) | -0.0918 (0.0738) | -0.103 (0.0685) | -0.107 (0.0818)
Statistical Analysis 1: Comparison: Group 1 (CC) vs Group 2 (NP2); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 52.1, 95% CI 2-sided [40.4 to 67.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 1 (CC) vs Group 3 (NP4); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 49.3, 95% CI 2-sided [39.0 to 62.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 1 (CC) vs Group 4 (NP8); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 40.8, 95% CI 2-sided [32.0 to 52.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1 (CC) vs Group 5 (NT); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 45.9, 95% CI 2-sided [35.7 to 59.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2 (NP2) vs Group 5 (NT); Test type: Superiority; p = 0.5817, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 113, 95% CI 2-sided [86.8 to 148] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3 (NP4) vs Group 5 (NT); Test type: Superiority; p = 0.8852, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 107, 95% CI 2-sided [83.7 to 138] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 4 (NP8) vs Group 5 (NT); Test type: Superiority; p = 0.6070, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 88.9, 95% CI 2-sided [68.7 to 115] — [estimate comment as in outcome 1, analysis 1]

17. Secondary Outcome: 3-OH-B[a]P Exposure in Subjects Using Nicotine Pouches for 7 Days Versus Subjects Who Continue to Smoke Cigarettes for 7 Days
Description: Summary of 24-hour urinary creatinine-adjusted 3-hydroxybenzo[a]pyrene (3-OH-B[a]P) in subjects using nicotine pouches (NP) for 7 days versus subjects who continue to smoke cigarettes for 7 days and subjects who stopped using any tobacco products for 7 days.
  Total urine weight (g) collected during 24 hours was converted to 24-hour urine volume using assumed density of 1 g = 1 mL
  Amount of biomarker was calculated as:
  Urine Biomarker (unit2/24 hours) = Urine biomarker concentration [unit1/mL] × 24h urine volume [mL] ÷ 1000, where: unit2 = ng if unit1 = pg; unit2 = μg if unit1 = ng
  Adjusted Urine biomarker (unit2/g creatinine) = Urine biomarker concentration (unit1/mL) × 100 / Creatinine concentration (mg/dL), where unit2 = ng if unit1 = pg, and unit2 = μg if unit 1 = ng
  The absolute change from baseline of urine biomarker amount excreted in 24 hours was calculated as follows:
  Absolute change from baseline = Post Randomization Value - Baseline Value
Time Frame: Samples collected over 24 hours on Day -1 (baseline) and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/g
Arm/Group | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
Number analyzed (Participants) | 28 | 22 | 30 | 25 | 21
pg/g
  Day -1 (Baseline) | 216 (155) | 139 (111) | 223 (158) | 172 (139) | 166 (101)
  Day 7 | 246 (215) | 30.8 (50.9) | 82.5 (105) | 57.7 (77.6) | 84.8 (174)
  Change from Baseline to Day 7 | 30.0 (192) | -108 (109) | -141 (186) | -115 (160) | -80.8 (195)
Statistical Analysis 1: Comparison: Group 1 (CC) vs Group 2 (NP2); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 13.2, 95% CI 2-sided [5.44 to 32.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 1 (CC) vs Group 3 (NP4); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 23.8, 95% CI 2-sided [10.7 to 53.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 1 (CC) vs Group 4 (NP8); Test type: Superiority; p = 0.0003, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 24.7, 95% CI 2-sided [10.6 to 57.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1 (CC) vs Group 5 (NT); Test type: Superiority; p = 0.0002, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 22.3, 95% CI 2-sided [9.21 to 54.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2 (NP2) vs Group 5 (NT); Test type: Superiority; p = 0.4280, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 59.1, 95% CI 2-sided [23.3 to 150] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3 (NP4) vs Group 5 (NT); Test type: Superiority; p = 0.9990, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 107, 95% CI 2-sided [44.8 to 255] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 4 (NP8) vs Group 5 (NT); Test type: Superiority; p = 0.9958, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 110, 95% CI 2-sided [44.9 to 272] — [estimate comment as in outcome 1, analysis 1]

18. Secondary Outcome: Urine Mutagenicity Exposure in Subjects Using Nicotine Pouches for 7 Days Versus Subjects Who Continue to Smoke Cigarettes for 7 Days
Description: Summary of 24-hour urine mutagenicity (Rev/24h) in subjects using nicotine pouches (NP) for 7 days versus subjects who continue to smoke cigarettes for 7 days and subjects who stopped using any tobacco products for 7 days.
  250 mL urine sample will be concentrated to 1 mL and used for urine mutagenicity testing.
  Measurement results are reported as revertants/μL. Urine mutagenicity count in the 24-hour urine was calculated as:
  Urine mutagenicity (revertants/250 mL) = Urine mutagenicity (revertants/μL) x 1000V, where V is the volume after concentration in mL
  Urine mutagenicity (revertants/24 hour) = Urine mutagenicity (revertants/250 mL) x [24h urine volume(mL) ÷ V], where V is the volume in mL of urine sample used for the mutagenicity test
Time Frame: Samples collected over 24 hours on Day -1 (baseline) and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Revertants / 24 hours
Arm/Group | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
Number analyzed (Participants) | 26 | 21 | 28 | 24 | 18
Revertants / 24 hours
  Day -1 (Baseline): number analyzed (Participants) | 26 | 20 | 28 | 24 | 18
  Day -1 (Baseline) | 13300 (14000) | 8770 (9480) | 9170 (11100) | 7580 (8210) | 12000 (12700)
  Day 7 | 10800 (13000) | 1710 (3150) | 2400 (3550) | 1920 (2440) | 3390 (5250)
  Change from Baseline to Day 7: number analyzed (Participants) | 26 | 20 | 28 | 24 | 18
  Change from Baseline to Day 7 | -2460 (8160) | -6980 (9170) | -6770 (11800) | -5650 (7460) | -8640 (9980)
Statistical Analysis 1: Comparison: Group 1 (CC) vs Group 2 (NP2); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means = -50.8, 95% CI 2-sided [-77.7 to -23.9] — Geometric least squares means were calculated by transforming the natural-log LS means back to the linear scale. Est. para. is ratio of geometric LS means for natural-log (expressed as a percentage), natural-log transformed back to the linear scale
Statistical Analysis 2: Comparison: Group 1 (CC) vs Group 3 (NP4); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means = -45.0, 95% CI 2-sided [-69.6 to -20.3] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 3: Comparison: Group 1 (CC) vs Group 4 (NP8); Test type: Superiority; p = 0.0003, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means = -42.3, 95% CI 2-sided [-68.2 to -16.5] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 4: Comparison: Group 1 (CC) vs Group 5 (NT); Test type: Superiority; p = 0.0004, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means = -44.8, 95% CI 2-sided [-72.6 to -17.0] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 5: Comparison: Group 2 (NP2) vs Group 5 (NT); Test type: Superiority; p = 0.9551, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means = -6.05, 95% CI 2-sided [-35.2 to 23.1] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 6: Comparison: Group 3 (NP4) vs Group 5 (NT); Test type: Superiority; p = 1.0000, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means = -0.198, 95% CI 2-sided [-27.3 to 26.9] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 7: Comparison: Group 4 (NP8) vs Group 5 (NT); Test type: Superiority; p = 0.9981, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means = 2.48, 95% CI 2-sided [-25.6 to 30.6] — [estimate comment as in outcome 18, analysis 1]

19. Secondary Outcome: 1-OH-Pyr Exposure in Subjects Using Nicotine Pouches for 7 Days Versus Subjects Who Continue to Smoke Cigarettes for 7 Days
Description: Summary of 24-hour urinary creatinine-adjusted 1-hydroxypyrene (1-OH-Pyr) in subjects using nicotine pouches (NP) for 7 days versus subjects who continue to smoke cigarettes for 7 days and subjects who stopped using any tobacco products for 7 days.
  Total urine weight (g) collected during 24 hours was converted to 24-hour urine volume using assumed density of 1 g = 1 mL
  Amount of biomarker was calculated as:
  Urine Biomarker (unit2/24 hours) = Urine biomarker concentration [unit1/mL] × 24h urine volume [mL] ÷ 1000, where: unit2 = ng if unit1 = pg; unit2 = μg if unit1 = ng
  Adjusted Urine biomarker (unit2/g creatinine) = Urine biomarker concentration (unit1/mL) × 100 / Creatinine concentration (mg/dL), where unit2 = ng if unit1 = pg, and unit2 = μg if unit 1 = ng
  The absolute change from baseline of urine biomarker amount excreted in 24 hours was calculated as follows:
  Absolute change from baseline = Post Randomization Value - Baseline Value
Time Frame: Samples collected over 24 hours on Day -1 (baseline) and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/g
Arm/Group | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
Number analyzed (Participants) | 28 | 22 | 30 | 25 | 21
μg/g
  Day -1 (Baseline) | 0.208 (0.147) | 0.148 (0.102) | 0.145 (0.0912) | 0.174 (0.114) | 0.174 (0.115)
  Day 7 | 0.198 (0.146) | 0.0489 (0.0485) | 0.0485 (0.0369) | 0.0506 (0.0372) | 0.0509 (0.0325)
  Change from Baseline to Day 7 | -0.00991 (0.102) | -0.0989 (0.0704) | -0.0969 (0.0817) | -0.123 (0.0822) | -0.123 (0.0935)
Statistical Analysis 1: Comparison: Group 1 (CC) vs Group 2 (NP2); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 31.7, 95% CI 2-sided [18.7 to 53.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Group 1 (CC) vs Group 3 (NP4); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 28.5, 95% CI 2-sided [17.6 to 46.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Group 1 (CC) vs Group 4 (NP8); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 24.3, 95% CI 2-sided [14.7 to 40.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Group 1 (CC) vs Group 5 (NT); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 28.1, 95% CI 2-sided [16.6 to 47.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Group 2 (NP2) vs Group 5 (NT); Test type: Superiority; p = 0.9511, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 113, 95% CI 2-sided [64.7 to 197] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Group 3 (NP4) vs Group 5 (NT); Test type: Superiority; p = 1.0000, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 101, 95% CI 2-sided [60.4 to 170] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Group 4 (NP8) vs Group 5 (NT); Test type: Superiority; p = 0.9003, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means (Test/Ref) = 86.5, 95% CI 2-sided [50.6 to 148] — [estimate comment as in outcome 1, analysis 1]

20. Secondary Outcome: Carboxyhemoglobin (COHb) Exposure in Subjects Using Nicotine Pouches for 7 Days Versus Subjects Who Continue to Smoke Cigarettes for 7 Days
Description: Summary of blood carboxyhemoglobin (%) in subjects using nicotine pouches (NP) for 7 days versus subjects who continue to smoke cigarettes for 7 days and subjects who stopped using any tobacco products for 7 days.
  The absolute change from baseline of urine biomarker amount excreted in 24 hours and blood biomarker concentration will be calculated as follows: Absolute change from baseline = Post Randomization Value - Baseline Value where Baseline = Day -1
Time Frame: Samples collected at approximately 21:30 on Day -1 (baseline) and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent saturation
Arm/Group | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
Number analyzed (Participants) | 26 | 21 | 28 | 24 | 18
percent saturation
  Day -1 (Baseline) | 11.8 (4.20) | 10.3 (3.59) | 11.3 (3.20) | 11.1 (5.25) | 11.0 (3.84)
  Day 7 | 11.3 (4.29) | 4.99 (1.67) | 4.60 (1.14) | 4.60 (0.918) | 4.22 (1.02)
  Change from Baseline to Day 7 | -0.585 (4.00) | -5.35 (4.01) | -6.65 (3.28) | -6.49 (5.12) | -6.77 (3.50)
Statistical Analysis 1: Comparison: Group 1 (CC) vs Group 2 (NP2); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means = 46.4, 95% CI 2-sided [37.1 to 58.0] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 2: Comparison: Group 1 (CC) vs Group 3 (NP4); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means = 43.1, 95% CI 2-sided [35.1 to 52.9] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 3: Comparison: Group 1 (CC) vs Group 4 (NP8); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means = 44.1, 95% CI 2-sided [35.5 to 54.6] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 4: Comparison: Group 1 (CC) vs Group 5 (NT); Test type: Superiority; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means = 39.1, 95% CI 2-sided [31.0 to 49.4] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 5: Comparison: Group 2 (NP2) vs Group 5 (NT); Test type: Superiority; p = 0.2351, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means = 119, 95% CI 2-sided [93.2 to 151] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 6: Comparison: Group 3 (NP4) vs Group 5 (NT); Test type: Superiority; p = 0.6570, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means = 110, 95% CI 2-sided [87.7 to 138] — [estimate comment as in outcome 18, analysis 1]
Statistical Analysis 7: Comparison: Group 4 (NP8) vs Group 5 (NT); Test type: Superiority; p = 0.5112, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio of geometric LS means = 113, 95% CI 2-sided [89.1 to 142] — [estimate comment as in outcome 18, analysis 1]

21. Secondary Outcome: Summary of Cigarettes Smoked Per Day (CPD)
Description: The number of cigarettes smoked per day (CPD) from 07:00 to 23:00 on Day 1 to Day 7 was collected to assess produce use behavior. Subjects in NP2, NP4, NP8 and NT groups were not allowed to use cigarettes starting at Day 1.
Time Frame: Data was collected from 07:00 to 23:00 each day starting from Day 1 to Day 7/end of study
Population: The Product Use Population includes all subjects from Groups 1, 2, 3, and 4 who used at least 1 of the assigned study products and all Group 5 subjects. Only subjects in the CC group were permitted to continue smoking their own brand of cigarettes and only data for these subjects is presented in the CPD summary.
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Group 1 (CC)
Number analyzed (Participants) | 29
cigarettes per day
  Day 1 | 16.1 (5.91)
  Day 2 | 15.8 (6.11)
  Day 3 | 15.6 (6.26)
  Day 4 | 14.8 (7.25)
  Day 5: number analyzed (Participants) | 28
  Day 5 | 15.8 (6.79)
  Day 6: number analyzed (Participants) | 28
  Day 6 | 15.8 (7.56)
  Day 7: number analyzed (Participants) | 28
  Day 7 | 15.9 (7.18)

22. Secondary Outcome: Summary of Total Number of Nicotine Pouches Used Per Day (NPPD)
Description: The number of nicotine pouches used per day (NPPD) from 07:00 to 23:00 on Day 1 to Day 7 was collected to assess produce use behavior. Only subjects in NP2, NP4 and NP8 groups used nicotine pouches during the study.
Time Frame: Data was collected from 07:00 to 23:00 each day starting from Day 1 to Day 7/end of study
Population: The Product Use Population includes all subjects from Groups 1, 2, 3, and 4 who used at least 1 of the assigned study products and all Group 5 subjects. Only subjects in NP2, NP4 and NP8 groups used nicotine pouch products during the study and data from only these subjects are provided in the NPPD summary.
Measure: Mean (Standard Deviation); unit: nicotine pouches per day
Arm/Group | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8)
Number analyzed (Participants) | 27 | 30 | 30
nicotine pouches per day
  Day 1 | 9.78 (6.00) | 9.77 (5.64) | 7.27 (4.96)
  Day 2: number analyzed (Participants) | 27 | 30 | 29
  Day 2 | 9.22 (6.16) | 10.2 (5.47) | 6.93 (4.06)
  Day 3: number analyzed (Participants) | 27 | 30 | 29
  Day 3 | 10.5 (7.12) | 9.87 (5.53) | 7.34 (4.56)
  Day 4: number analyzed (Participants) | 27 | 30 | 27
  Day 4 | 9.48 (6.46) | 10.2 (6.25) | 7.15 (4.00)
  Day 5: number analyzed (Participants) | 25 | 30 | 25
  Day 5 | 10.1 (6.82) | 10.4 (5.70) | 7.36 (4.24)
  Day 6: number analyzed (Participants) | 25 | 30 | 25
  Day 6 | 10.7 (6.34) | 10.1 (5.71) | 7.12 (3.88)
  Day 7: number analyzed (Participants) | 24 | 30 | 25
  Day 7 | 10.8 (7.77) | 11.2 (6.91) | 7.60 (4.24)

23. Secondary Outcome: Summary of Average Number of Nicotine Pouches Per Use
Description: The average number of nicotine pouches per use occasion (NPPU) from 07:00 to 23:00 on Day 1 to Day 7 was collected to assess produce use behavior. Only subjects in NP2, NP4 and NP8 groups used nicotine pouches during the study.
Time Frame: Data was collected from 07:00 to 23:00 each day starting from Day 1 to Day 7/end of study
Population: The Product Use Population includes all subjects from Groups 1, 2, 3, and 4 who used at least 1 of the assigned study products and all Group 5 subjects. Only subjects in NP2, NP4 and NP8 groups used nicotine pouch products during the study and data from only these subjects are provided in the NPPU summary.
Measure: Mean (Standard Deviation); unit: nicotine pouches per use
Arm/Group | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8)
Number analyzed (Participants) | 27 | 30 | 30
nicotine pouches per use
  Day 1 | 1.19 (0.309) | 1.22 (0.285) | 1.09 (0.204)
  Day 2: number analyzed (Participants) | 27 | 30 | 29
  Day 2 | 1.22 (0.434) | 1.28 (0.404) | 1.15 (0.378)
  Day 3: number analyzed (Participants) | 27 | 30 | 29
  Day 3 | 1.26 (0.468) | 1.33 (0.575) | 1.21 (0.444)
  Day 4: number analyzed (Participants) | 27 | 30 | 27
  Day 4 | 1.25 (0.436) | 1.32 (0.389) | 1.18 (0.308)
  Day 5: number analyzed (Participants) | 25 | 30 | 25
  Day 5 | 1.26 (0.420) | 1.33 (0.419) | 1.13 (0.255)
  Day 6: number analyzed (Participants) | 25 | 30 | 25
  Day 6 | 1.35 (0.461) | 1.35 (0.481) | 1.13 (0.256)
  Day 7: number analyzed (Participants) | 24 | 30 | 30
  Day 7 | 1.37 (0.513) | 1.38 (0.473) | 1.13 (0.227)

24. Secondary Outcome: Summary of Average Duration of Each Nicotine Pouch Use
Description: The average duration (in minutes) of each nicotine pouch use from 07:00 to 23:00 on Day 1 to Day 7 was collected to assess produce use behavior. Only subjects in NP2, NP4 and NP8 groups used nicotine pouches during the study.
Time Frame: Data was collected from 07:00 to 23:00 each day starting from Day 1 to Day 7/end of study
Population: The Product Use Population includes all subjects from Groups 1, 2, 3, and 4 who used at least 1 of the assigned study products and all Group 5 subjects. Only subjects in NP2, NP4 and NP8 groups used nicotine pouch products during the study and data from only these subjects are provided in the summary for average duration of each nicotine pouch use.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8)
Number analyzed (Participants) | 27 | 30 | 30
minutes
  Day 1 | 23.5 (13.3) | 22.4 (10.3) | 19.1 (11.4)
  Day 2: number analyzed (Participants) | 27 | 30 | 29
  Day 2 | 25.1 (11.8) | 25.1 (13.2) | 21.6 (13.6)
  Day 3: number analyzed (Participants) | 27 | 30 | 29
  Day 3 | 27.6 (13.4) | 25.5 (14.5) | 23.3 (13.5)
  Day 4: number analyzed (Participants) | 27 | 30 | 27
  Day 4 | 27.6 (15.1) | 25.4 (11.0) | 26.2 (18.5)
  Day 5: number analyzed (Participants) | 25 | 30 | 25
  Day 5 | 27.4 (14.2) | 27.3 (13.2) | 26.8 (18.8)
  Day 6: number analyzed (Participants) | 25 | 30 | 25
  Day 6 | 30.1 (13.8) | 26.0 (13.1) | 28.9 (20.2)
  Day 7: number analyzed (Participants) | 24 | 30 | 25
  Day 7 | 25.5 (13.0) | 24.5 (12.4) | 27.3 (19.7)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from the time the subject first signs the ICF (within 28 days prior to randomization) to final discharge from the study (up to 8 days after randomization).
Description: Subjects were observed for any signs or symptoms and asked about their condition by open questioning, such as "How have you been feeling since you were last asked?", at least once each day while resident at the study site and at each study visit. Subjects were also be encouraged to spontaneously report AEs occurring at any other time during the study.
Arm/Group | Not Assigned | Group 1 (CC) | Group 2 (NP2) | Group 3 (NP4) | Group 4 (NP8) | Group 5 (NT)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/29 | 0/28 | 0/30 | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/29 | 0/28 | 0/30 | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 0/2 | 5/29 | 15/28 | 9/30 | 15/30 | 12/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Not Assigned (N=2) | Group 1 (CC) (N=29) | Group 2 (NP2) (N=28) | Group 3 (NP4) (N=30) | Group 4 (NP8) (N=30) | Group 5 (NT) (N=29)
Headache (Nervous system disorders) | 0 | 4 | 6 | 5 | 4 | 4
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gingival discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lip disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol: ALCS-REG-20-15-OTDN Protocol Version 3 (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT05664672/Prot_000.pdf
  • Study Protocol: ALCS-REG-20-15-OTDN Protocol Version 2 (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/72/NCT05664672/Prot_001.pdf
  • Study Protocol: ALCS-REG-20-15-OTDN Protocol Version 1 (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT05664672/Prot_002.pdf
  • Statistical Analysis Plan (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT05664672/SAP_003.pdf